CLINICAL TRIAL: NCT04003415
Title: Respiratory Disorders Non-invasive Monitoring of Work of Breathing in Outpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Work of Breathing Study Group (Unknown)
Responsible Party: Principal Investigator, Andrea Jonas, Pulmonary & Critical Care Fellow, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB-51805
Record Dates: First submitted 2019-06-26; First posted 2019-07-01 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Copd; Asthma; Respiratory Effort; Contactless Vital Sign Monitoring
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma | interventions — Heart Rate; Electrocardiography; Monitoring, Physiologic; Oximetry

STUDY DESIGN:
Intervention Model Description: All participants enrolled in the study will be in the intervention arm. Intervention consists of device feasibility and validation of heart rate and respiratory rate data collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Investigational Device Arm (Experimental): Once consented for the study, participants will undergo testing with the investigational device for a one hour period. Testing will entail the participant wearing an EKG monitor, a respiratory rate monitor, a pulse oximeter, and being positioned next to the investigational device. The investigational device is contactless and captures chest movement of participants which allows it to estimate real time heart rate and respiratory rate. Additional data collected with the EKG monitor, respiratory rate monitor, and the pulse oximeter will be used to validate the vital sign data collected by the investigational device. After data collection is complete, participant involvement will then be over. Participants will have the option to return on a later date for additional testing (up to a maximum of three sessions total), within the six month window of the study. Participants will continue their standard of care therapies for their respiratory condition.
  Interventions: Device: Investigational Device: Contactless heart rate and respiratory rate monitor; Diagnostic Test: Heart Rate (EKG) Monitor; Diagnostic Test: Respiratory rate Monitor; Diagnostic Test: Pulse Oximetry

INTERVENTIONS:
Device: Investigational Device: Contactless heart rate and respiratory rate monitor — Participant will be seated next to the investigational device. The device is contactless, and will measure the patient's heart rate and respiratory rate through use of radio-waves.
  Other Names: Investigational Device
Diagnostic Test: Heart Rate (EKG) Monitor — Participant will undergo 3-lead EKG testing to measure heart rate during testing.
Diagnostic Test: Respiratory rate Monitor — Participant will have an elastic band around their chest for monitoring respiratory rate during testing.
Diagnostic Test: Pulse Oximetry — Participants will wear a finger pulse oximeter during the testing for monitoring of heart rate, respiratory rate, and pulse oximetry.

SUMMARY:
This study will test the accuracy of an investigational, non-invasive device for measuring heart rate and respiratory rate. The device emits radiowaves that allows it to pick up subtle changes in a person's chest wall, which allows it to calculate the heart rate and respiratory rate. We propose to study whether the device's measurements are accurate and reproducible in patients with chronic obstructive pulmonary disease (COPD) or asthma. The device undergoing study has been evaluated in healthy volunteers, but its accuracy in vital sign monitoring in patients with respiratory conditions has not yet been established. This study will serve as the foundation for additional work to assess the device's accuracy in measuring a patient's overall "work of breathing" or respiratory effort. Future work will examine the device's accuracy in measuring work of breathing in patients having an exacerbation of their underlying respiratory condition.

The primary aim of this study will be to assess the validity of heart rate and respiratory rate measurements in patients with either COPD or asthma.

ELIGIBILITY:
Inclusion Criteria:

* Patient seen at the Stanford University Hospital Chest Clinic
* Patient age 18 or older
* Patient able to consent
* Patient with one of the following two medical conditions: Chronic Obstructive Pulmonary - Disease or Asthma
* Participant (or accompanying family / caretaker) able to speak English

Exclusion Criteria:

* Patient does not meet inclusion criteria (under age 18, unable to consent, etc.)
* Patient is hospitalized
* Patient is having an acute exacerbation of their respiratory condition
* Patient is having an acute exacerbation of a comorbid condition
* Patient has comorbid cardiac disease, including one of the conditions listed below:
* Arrhythmias (including atrial fibrillation, NSVT, etc.)
* Congestive Heart Failure
* Unstable angina
* Myocardial infarction within the last 3 months prior to enrollment
* Uncorrected congenital heart disease
* Uncorrected severe valvular disease
* Pulmonary Hypertension (moderate or higher grade)
* Patient has one of the following conditions:
* Moderate pleural effusion
* Large pleural effusion
* Advanced stage lung cancer (Stage III or Stage IV disease)
* Active infectious process, including viral process or pneumonia
* Interstitial lung disease
* Pleural disease, including pleural malignancies, trapped lung, etc
* Active Cheyne-Stokes respiration
* Patient has baseline increased work of breathing not due to their underlying respiratory disease (ie. COPD or asthma)
* Ongoing substance abuse (not including cigarette use)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Heart Rate | 30 - 60 minutes
  Heart rate data as compared between the investigational device, a 3-lead EKG, and a finger probe.
Respiratory rate | 30 - 60 minutes
  Respiratory rate data as compared between the investigational device, a respiratory rate monitor, and a finger probe.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Jonas, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Full Access: Access to Data, Access to patient PHI, Access to RedCap Document linking patients to their study numbers.
  Limited Access: Access to de-identified participant data for analysis
  Study PI and Study Faculty Sponsor: Full Access Research Team and Industry Sponsors: Limited Access
  Upon enrollment each participant will be assigned a unique study number. Any study data collected will be linked to the patient solely through the study number. The document that contains the patient information and their study numbers will by kept on Stanford RedCap and will only be accessible by the study PI and the faculty sponsor. De-identified data of vital sign measurements will be shared between the Stanford research team and industry collaborators. Data will be downloaded to an encrypted USB key and hand-delivered between members of the research team. For smaller files, de-identified patient data will be mailed securely between the research team members.
Supporting Information: Study Protocol, SAP
Time Frame: Data collection will take place over the course of a 6 month period. De-identified patient data will be kept for a period of 5 years.
Access Criteria: Access to patient PHI will be limited to the study PI and the faculty sponsor. Access to de-identified patient data will be allowed for research and industry collaborators for analysis.

REFERENCES:
- [Background] W. Li, B. Tan and R. J. Piechocki,
- [Background] Levitas, I. Naidionova and J. Matuzas,
- See also: Reference 1 — http://ieeexplore.ieee.org/stamp/stamp.jsp?tp=&arnumber=7511389&isnumber=7510595
- See also: Reference 2 — http://ieeexplore.ieee.org/stamp/stamp.jsp?tp=&arnumber=6869188&isnumber=6869176